CLINICAL TRIAL: NCT02334696
Title: Improving Outcomes in Vascular Access
Acronym: IMPROVA
Status: Terminated | Type: Observational
Why Stopped: similar study in USA published with same protocol
Sponsor: University Hospital Birmingham (Other)
Responsible Party: Principal Investigator, Mr Nick Inston, Renal Surgery Consultant, University Hospital Birmingham
Other Study IDs: RRK5258
Record Dates: First submitted 2015-01-06; First posted 2015-01-08 (Estimated); Last update posted 2019-04-26 (Actual); Status verified 2019-04

CONDITIONS: End Stage Renal Disease
Keywords: Vascular Access
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The IMPROVA study is designed to identify novel predictors of vascular access success or failure. Clinical assessment complimented by Doppler ultrasound is the only currently employed methods of assessing suitability for placement of arteriovenous fistulae (AVF). These techniques are not capable of predicting vascular access outcomes suggesting that other potentially measurable factors may play a part.

Despite efforts to improve placement of AVF in both the haemodialysis incident and prevalent population, many patients continue to dialyse through a central venous catheter (CVC), exposing them to higher risks of infection, co morbidity and mortality than dialysing via an AVF. Furthermore, AVF primary failure rates are reportedly as high in 20-50% in published series confirming that ultrasound cannot inform the clinician sufficiently to accurately predict success or failure.

The aim of this study is to perform enhanced assessments of arterial health preoperatively and correlate these measurements with early AVF outcome. We intend to perform pulse wave analysis and velocity; measure advanced glycation end products and assess endothelial function using a vascular occlusion test. We also aim to assess whether patient reported symptoms of hand function can predict AVF outcome. These non-invasive measurements will provide a more accurate picture of overall vascular health prior to AVF formation with the ultimate intention of informing the clinician as to the likelihood of success or failure.

DETAILED DESCRIPTION:
Purpose of proposed investigation The IMPROVA study will utilise novel non-invasive methods of arterial health assessment and correlate these measurements with the early outcomes of AVF formation. The development of new techniques to inform the clinician pre-operatively will aid in a more tailored approach to fistula planning, predict inevitable failures and consequently improve success rate. The ultimate aim is to identify novel methods of predicting fistula failure to prevent patients from developing into a cycle of consecutive failure, catheter dependence and therefore worse overall outcomes.

Background Despite the merits of autologous arteriovenous fistulas (AVF), failure rates remain high with 20-50% failing to mature. As a consequence many patients will suffer multiple attempts at establishing arteriovenous access and initiate dialysis on a Central Venous Catheter (CVC) thereby extending this risk of subsequent failure and increasing the risk of mortality and serious comorbidity.

Predictors of maturation have been reported in a number of studies. The mainstay is pre-operative vascular mapping by duplex ultrasonography (DUS) which relies on vessel size and site. Whilst this has demonstrated improved patency and decreased early failure rate vascular measurements are unable to independently predict outcome of fistula success suggesting other contributing factors.

The process of maturation can be modelled around changes in blood flow, flow patterns and subsequent vessel dilatation and remodelling. The ability of the artery and vein to dilate is essential to fistula maturation.

Factors that influence vessel remodelling following fistula formation have been under investigated in this important aspect in the management of kidney disease. Arterial stiffness refers to the distensability, compliance and elastic modulus of the arterial vascular system. It is found to increase with age, diabetes mellitus, atherosclerosis and end stage renal disease. Aortic pulse wave velocity is considered the gold standard for assessing arterial stiffness and the pulse wave Vicorder©Skidmore Medical is a non-invasive, easy to learn and reproducible method of assessing stiffness. Increased aortic pulse wave velocity has been independently associated with adverse cardiovascular outcome in large prospective studies including specifically patients with end stage renal failure. Advanced glycation end products (AGEs) have also been implicated in the development of vascular pathology resulting in AVF failure. The measurement of advanced glycation end products, using the AGE reader©Diagnoptics Technologies, offers a new avenue to establish the association between AGE levels and AVF outcomes. Furthermore, potential therapeutic options exist for improving the AGE-related vascular biology of AVFs with evidence that aminoguanine, ALT-946, ALT-711, statins, pyrodoxamine and dietary modifications can reduce AGE levels. Endothelial function is another aspect of arterial health that has been under reported in vascular access research. The INVOS® spectra machine uses near infrared spectroscopy to measure the mixed arteriovenous saturations of deep tissues as a reflection of perfusion. Manipulation of this environment using a vascular occlusion test can provide invaluable information regarding endothelial responsiveness. Patient reported symptoms of vascular health may also provide important information in the search for novel predictors of AVF outcomes. Many vascular diseases have associated symptoms that reflect severity and direct questioning of patients regarding the vascular health of their upper limbs may offer further guidance in the placement of AVF.

The combination of these non-invasive, easy to learn and reproducible tests offers an exciting opportunity to identify predictors of and improve outcomes in AVF formation.

ELIGIBILITY:
Inclusion Criteria:

Age 18 years or more. All patients referred to the vascular access clinic. Able to give valid informed consent.

Exclusion criteria Unable to give informed consent. <18 years old Prisoners

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with end stage renal disease referred for assessment in vascular access clinic.
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2015-01; Primary Completion 2016-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Early patency | 2 - 6 weeks
  A successful fistula is defined as any fistula which at early postoperative review shows:
  Fistula flow rates >600ml/min Fistula vein diameter >6mm Distance of fistula vein from skin <6mm
  - 10% allowable for flow rates and vein diameter A failed fistula is defined as any fistula which does not meet this definition.

SECONDARY OUTCOMES:
Unassisted clinical maturation | 12 months
  Use of fistula with 2 needles for 75% of dialysis sessions during a 4-wk period with either:
  1. 4 consecutive dialysis sessions with mean blood pump speed >300 mL/min, or
  2. single-pool Kt/V >1.4 or urea reduction ratio >70%